CLINICAL TRIAL: NCT06792643
Title: Efficacy and Safety of Cangrelor on Top of anticoagUlation in Patients With myocaRdial Infarction Related Cardiogenic Shock/Cardiac Arrest receiVIng VAECMO Support - a Phase 2, Single Arm, Single Center Trial
Brief Title: Cangrelor on Top of anticoagUlation in Patients With myocaRdial Infarction-related Cardiogenic Shock/Cardiac Arrest receiVIng VA-ECMO
Acronym: SURVIVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Anna Mara Scandroglio, Principal Investigator, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURVIVE
Record Dates: First submitted 2023-10-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation Complication; Platelet Dysfunction
Keywords: Cangrelor; ACS; Cardiogenic Shock; PCI; ECMO; VA-EMO; Acute coronary syndrome; P2Y12; Anti-thrombotic therapy; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Shock, Cardiogenic; Acute Coronary Syndrome | interventions — cangrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cangrelor (Experimental): Cangrelor will be started without bolus at a low dose of 0.125 mcg/kg/min and titrated (by 0.125 mcg/kg/min steps) based on the results of platelet function assay to guarantee effective platelet P2Y12 pathway inhibition.
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Cangrelor — Cangrelor will be started without bolus at a low dose of 0.125 mcg/kg/min and titrated (by 0.125 mcg/kg/min steps) based on the results of platelet function assay to guarantee effective platelet P2Y12 pathway inhibition.

SUMMARY:
The SURVIVE trial aims to test whether using an anti-thrombotic regimen involving cangrelor can reduce bleeding risk while maintaining effective antithrombotic effects in patients on VA-ECMO due to cardiogenic shock (CS)/ cardiac arrest (CA) who undergo percutaneous coronary intervention (PCI). The investigators plan to achieve this by starting cangrelor on top of systemic anticoagulation with bivalirudin at a low dose, regularly monitoring platelet function, and adjusting the dose based on the results of platelet function assay (Multiplate®) to guarantee effective platelet P2Y12 pathway inhibition to achieve optimal platelet inhibition. Platelet function assays will be performed at various time points throughout the treatment timeframe. Cangrelor will then be stopped at the end of VA-ECMO support, and patients will be transitioned to oral P2Y12- inhibitors as per clinical guidelines.

DETAILED DESCRIPTION:
Veno-Arterial Extra Corporeal Membrane Oxygenation (VA-ECMO) is increasingly used to support patients throughout a spectrum of hemodynamic instability states ranging from severe cardiogenic shock (CS) to refractory cardiac arrest (CA). VA-ECMO, is thus often employed in clinical practice for the management of CS/CA complicating acute coronary syndromes (ACS). The interface of blood and VA-ECMO mechanical components, along with rotational forces generated by pump impellers configures a unique combination of prothrombotic and pro-haemorrhagic milieu (haemocompatibility). In this setting of competing thrombotic and hemorrhagic risks, optimal anti-thrombotic therapy remains ill-defined for patients undergoing percutaneous coronary intervention (PCI) for ACS on VA-ECMO. Theoretically, dual anti-platelet therapy (DAPT) consisting of aspirin plus an oral P2Y12 inhibitor should be associated with systemic anticoagulation (triple antithrombotic therapy). Platelet activation during ECMO support confers increased thrombotic risk, which, in the setting of ACS-related CS/CA, is worsened by the pro-thrombotic and pro-inflammatory state, the low-cardiac output with subsequent blood stasis and tissue hypoperfusion and possibly the need for myocardial revascularization procedure with stent implantation. At the same time, blood interaction with device foreign surfaces has been associated to reduced platelet surface expression of GpIb-GpIV, lower activated surface GpIIb-IIIa levels and blunted ADP-mediated aggregation, which translate into increased bleeding risk. Bleeding complications, however, exceed ischemic risk and triple antithrombotic therapy may confer an excess risk in this population prone to bleeding and may jeopardize patients' outcome. In this context of delicate haemostatic equilibrium several pharmacokinetic and pharmacodynamic factors limit the use of standard DAPT in addition to systemic anticoagulation, including the irreversible inhibiting effect of aspirin on platelets and the relatively long duration of action of oral P2Y12 inhibitors.

In addition, while GpIIb-IIIa inhibitors may offer a parenteral alternative antiplatelet agent, their use has been associated with increased transfusion need during VA-ECMO. The study hypothesis is that an anti-thrombotic regimen comprising cangrelor, an intravenous non-thienopyridine, reversible adenosine-diphosphate P2Y12 receptor antagonist, may reduce bleeding risk while providing adequate antithrombotic effect in patients on VA ECMO due to CS/CA who underwent PCI. Both the rapid onset and offset of action of this agent make it a particularly attractive option in patients at a high risk of both thrombotic and haemorrhagic complications, since a combination of a low starting dose of cangrelor coupled with regular platelet function tests potentially guarantees achieving adequate anti-platelet effect at the lowest possible cangrelor dose, in order to prevent ischemic events while minimizing bleeding risk.

Systemic anticoagulation will be performed with bivalirudin, titrated to achieve effective systemic anticoagulation and an activated thromboplastin time (aPTT) of 55-70'', as for routine clinical practice. Cangrelor will be started without bolus at a low dose of 0.125 mcg/kg/min and titrated (by 0.125 mcg/kg/min steps) based on the results of platelet function assay to guarantee effective platelet P2Y12 pathway inhibition. Platelet function will be assessed with the Multiplate analyser with the aim to reach and ADP-test <46 U. Platelet assay will be performed at baseline, 30 min after cangrelor infusion start, 12 hours after cangrelor infusion start, after any cangrelor dose modulation, regularly every 24 hours, at time of any thrombotic/bleeding event, and up to 48 hours from oral P2Y12-inhibitor initiation. Treatment with cangrelor will be discontinued at the end of VA-ECMO support, and patients will be loaded with oral P2Y12-inhibitors, as recommended for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years;
* ACS-related CS/CA patients undergoing PCI (either with or without stent implantation) and needing VA-ECMO support;
* Patients who received pre-hospital aspirin intravenous loading dose or patients naïve to any anti-thrombotic agent;
* Written informed consent

Exclusion Criteria:

* Overt uncontrollable bleeding;
* Suspected intra-cranial haemorrhage;
* Patients who received any dose of any oral P2Y12-inhibitors;
* Patients with known history of stroke or Transient Ischaemic Attack (TIA);
* Patients with known hypersensitivity to the active substance (cangrelor) or to any of its excipients;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major bleeding [type 3b or 5 Bleeding Academic Research Consortium (BARC) bleeding] - Safety outcome | Up to 48 hours after ECMO support withdrawal
  Major bleeding will be defined as type 3b or 5 Bleeding Academic Research Consortium (BARC) bleeding.
Thrombotic events - Efficacy outcome | Up to 48 hours after ECMO support withdrawal
  Thrombotic events will be defined as: any new myocardial infarction, any definite or probable stent thrombosis (ST) according to Academic Research Consortium (ARC)-2 criteria, any peripheral arterial thrombosis, any venous thrombosis/venous thromboembolism or imaging-defined ischemic stroke.
Multiplate assay with ADP-test values <46 U | Up to 48 hours after ECMO support withdrawal
  Multiplate assay with ADP-test values <46 U (time in therapeutic range)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request after approval of the PI.